CLINICAL TRIAL: NCT03967392
Title: Comparison of Bupivacaine Versus Bupivacaine-dexamethasone Infiltration for Postoperative Analgesia in Skin Graft Donor Sites, a Randomized Trial
Brief Title: Comparison of Bupivacaine Versus Bupivacaine-dexamethasone Infiltration for Postoperative Analgesia in Skin Graft Donor Sites
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, RAMY AHMED, lecturer of anesthesia at faculty of medicine ain shams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ain Shams UNIVER
Record Dates: First submitted 2019-05-22; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Postoperative Pain Atskin Graft Site
Keywords: Bupivacaine,dexamethasone,Analgesia,Skin Graft ,Donor
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: DOUBLE BLINDED RANDOMELY CONTROLLED
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP X(xylocaine) (Active Comparator): 20 ml bupivacaine 0.5% + 20 ml normal saline.
  Interventions: Drug: Xylocaine
- GROUPX(Dxylocaine and dexamethasone) (Active Comparator): 20 ml bupivacaine 0.5% + 18 ml normal saline + 8 mg dexamethasone 2 ml
  Interventions: Drug: Xylocaine

INTERVENTIONS:
Drug: Xylocaine — TREATMENT

SUMMARY:
Background: Skin grafting; both partial and complete thickness is frequently used in reconstruction of traumatic soft tissue defects. It is of great value not only for functional and aesthetic purposes in the field of plastic surgery, but also for other surgical specialties.

Of all the problems in the early postoperative period, pain is considered the most important, ameliorating it can lead to significant reduction in postoperative morbidity and faster recovery of the skin donor site.

Objective: To evaluate use of dexamethasone as adjuvant for bupivacaine in subcutaneous local anesthesia infiltration for skin graft donor sites, on quality of pain relief and total dose of analgesic requirements in the early hours postoperatively.

Methods: 97 patients were randomly allocated to receive local bupivacaine infiltration (group LB), or dexamethasone plus bupivacaine (group LB + D) in skin donor site after skin harvesting. In addition to basic demographic data; patients were compared for Numerical Rating Scale (NRS), total dose of morphine or morphine equivalents, time to 1st breakthrough pain, and duration of surgery.

Keywords: Donor site. skin graft. Breakthrough pain. Rescue analgesia. Bupivacaine

DETAILED DESCRIPTION:
The patients included in the study were randomly allocated to 1 of 2 parallel groups: 1) bupivacaine plus dexamethasone (LB+D) group (n = 50): received 20 ml bupivacaine 0.5% + 18 ml normal saline + 8 mg dexamethasone 2 ml, 2) bupivacaine only (LB) group (n = 50): received 20 ml bupivacaine 0.5% + 20 ml normal saline. A random allocation sequence was generated electronically using online randomization service from https://www.random.org. The project medicine was prepared by 2 independent assistants not involved in other parts of the study. All persons involved were blinded to the randomized allocation.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists Physical Status classification I-II and scheduled for split thickness skin grafting to cover full thickness skin burn or degloving injury after trauma.

Exclusion Criteria:

* were inability to cooperate.
* immunosuppressive therapy.
* Body Mass Index > 35.
* diabetes.
* lower-limb neuropathy.
* daily intake of glucocorticoids or opioids.
* patients who need area of coverage more than 10 cm2.
* allergy to any drug used in the study.
* alcohol or drug abuse.
* American Society of Anesthesiologists Physical Status classification III or more.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-75 YEARS
Enrollment: 100 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
Numeric Rating scale for pain assesment during the first postoperative 12 hours | 4 MONTHS
  TREATMENT

CONTACTS AND LOCATIONS:
Locations (1):
- Ramymahrose, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No